CLINICAL TRIAL: NCT00102869
Title: Dopaminergic Enhancement of Learning and Memory (LL_001, Project on Aphasia)
Brief Title: Dopaminergic Enhancement of Learning and Memory in Aphasia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Rainer Girgenrath, Bundesministerium für Bildung und Forschung (BMBF)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LL_001, Project on aphasia
Record Dates: First submitted 2005-02-03; First posted 2005-02-04 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2008-06

CONDITIONS: Cerebrovascular Accident; Aphasia
Keywords: language acquisition; plasticity; stroke recovery; aphasia treatment; naming; levodopa; stroke
MeSH Terms: conditions — Stroke; Aphasia | interventions — Levodopa

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: levodopa — 100mg levodopa per day over 10 days/ treatment phase

SUMMARY:
The purpose of this study is to determine whether levodopa, in combination with a high frequency language training, is effective in boosting naming performance in patients with aphasia.

DETAILED DESCRIPTION:
Our prior work shows that d-amphetamine and the dopamine precursor levodopa markedly improve word learning success in healthy subjects. In this randomized, placebo-controlled, double-blind clinical trial, we probe whether daily administration of levodopa, coupled with several hours of language training every day, will significantly improve naming abilities in patients with aphasia as compared to placebo administration. We furthermore examine with magnetic resonance imaging which brain regions need to be functionally intact for a dopaminergic improvement of language therapy.

ELIGIBILITY:
Inclusion Criteria for patients with aphasia:

* Unilateral cerebrovascular accident (stroke) in the territory of the arteria media
* Time post onset: > 6 months
* Aphasia with anomia
* Age between 18-75 years
* Premorbid right-handedness
* Primary language: German

Exclusion Criteria for patients and healthy controls:

* Known allergy to levodopa or tartrazine
* History of medication/drug abuse
* Acute nicotine withdrawal or > 15 cigarettes per day
* > 6 cups/glasses of coffee, caffeine drinks or energy drinks per day
* > 50 grams of alcohol per day
* Severe hypertonia (systole >180 mm Hg)
* Severe arteriosclerosis
* Diabetes, asthma, or glaucoma
* Severe hearing disability
* Evidence for severe hippocampal damage
* Premorbid depression or psychosis
* Medication with dopamine agonists or antagonists
* Parkinsonian symptoms
* Changes in anticonvulsive medication during the week prior to study enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-01; Primary Completion 2007-02 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Boost in naming performance (percent correct) through levodopa as compared to placebo | immediately after each treatmentphase
Brain activity pattern in successfully trained patients | immediately after each treatmentphase

SECONDARY OUTCOMES:
Stability of naming performance after one month and six months post treatment | from 1 month untill 6 months after treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Breitenstein, PhD, Study Director — Dept. of Neurology, University Hospital Muenster, Germany; Stefan Knecht, MD, Study Chair — Dept. of Neurology, University Hospital Muenster, Germany
Locations (1):
- Dept. of Neurology, University Hospital Muenster, Münster, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Knecht S, Breitenstein C, Bushuven S, Wailke S, Kamping S, Floel A, Zwitserlood P, Ringelstein EB. Levodopa: faster and better word learning in normal humans. Ann Neurol. 2004 Jul;56(1):20-6. doi: 10.1002/ana.20125. PMID 15236398
- [Background] Breitenstein C, Wailke S, Bushuven S, Kamping S, Zwitserlood P, Ringelstein EB, Knecht S. D-amphetamine boosts language learning independent of its cardiovascular and motor arousing effects. Neuropsychopharmacology. 2004 Sep;29(9):1704-14. doi: 10.1038/sj.npp.1300464. PMID 15114342
- [Background] Breitenstein C, Knecht S. [Language acquisition and statistical learning]. Nervenarzt. 2003 Feb;74(2):133-43. doi: 10.1007/s00115-002-1466-1. German. PMID 12596014
- [Derived] Breitenstein C, Korsukewitz C, Baumgartner A, Floel A, Zwitserlood P, Dobel C, Knecht S. L-dopa does not add to the success of high-intensity language training in aphasia. Restor Neurol Neurosci. 2015;33(2):115-20. doi: 10.3233/RNN-140435. PMID 25588456